CLINICAL TRIAL: NCT05186480
Title: Evaluation of the Effect of Immune Modulating Enteral Nutrition Formula Versus Regular Enteral Nutrition on the Outcome of Critically Ill Sepsis Patients. A Pilot Study
Brief Title: Evaluation of the Effect of Immune Modulating Enteral Nutrition Formula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NewGiza University (Other)
Responsible Party: Principal Investigator, Rana Muhammed, Principle Investigator, NewGiza University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NewGizaU
Record Dates: First submitted 2021-10-28; First posted 2022-01-11 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Sepsis; Critical Illness
Keywords: malnutrition; immune modulating formula
MeSH Terms: conditions — Sepsis; Critical Illness; Malnutrition

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Active Comparator): they receive the immune enhancing formula
  Interventions: Dietary Supplement: Neo Mune
- control group (No Intervention): they receive the conventional formula

INTERVENTIONS:
Dietary Supplement: Neo Mune — Neo-mune is a nutritional formula used in enteral feeding for critically ill patients. It's mainly indicated in cases of malnutrition, post surgeries and traumas and immunocompromisation.
  Its composition:
  Composition in approximate %w/w Maltodextrin 42.44% Sodium caseinate 18.25% MCT oil 6.28% Arginine 5.21% Polydextrose 4.00% Corn oil 3.48% Glutamine 2.61% Fish oil 2.32% Minerals 1.96% Vitamins 0.86% Artificial flavor (vanilla)
  Arms: test group

SUMMARY:
The aim is to compare the efficacy and tolerability of an immune modulating enteral nutrition formula versus the regular formula on the outcomes of critically ill septic patients by assessment of clinical outcomes, immune profile, tolerability and enteral nutrition intolerance and laboratory markers

DETAILED DESCRIPTION:
Nutritional formulas are considered important sources of the dietary components that the body requires. They contain the sources of fats, proteins and carbohydrates and compensate any vitamin and mineral deficiency.

There is a special type of formulas called the "immune-enhancing formulas", they supplement the body not only with the energy sources but also, they boost the body's immune system as they contain multiple types of amino and fatty acids.

There is an ongoing debate around the efficacy of the immune-enhancing formulas, some studies show that they make a significant difference in enhancing the clinical outcomes compared to traditional formulas while other studies showed no significant difference between the traditional formulas and immune-enhancing formula.

The immune-enhancing nutritional formula is used in enteral and oral feeding for critically ill patients. It's mainly indicated in cases of malnutrition, post surgeries and traumas and immunocompromised patients.

Its composition:

Composition in approximate %w/w Maltodextrin 42.44% Sodium caseinate 18.25% MCT oil 6.28% Arginine 5.21% Poly-dextrose 4.00% Corn oil 3.48% Glutamine 2.61% Fish oil 2.32% Minerals 1.96% Vitamins 0.86% Artificial flavor (vanilla)

This study analyzed prospectively the clinical and laboratory outcomes of critically ill sepsis patients taking regular enteral nutrition versus immune modulating formulas.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with sepsis according to guideline criteria AND
* Age ≥18 years

Exclusion Criteria:

* Gastrointestinal tract complications or intestinal failure or any contraindications to receive enteral nutrition
* Hemodynamic instability on admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-03 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-28 (Estimated)

PRIMARY OUTCOMES:
Intensive Care Unit mortality | 28 days
  The Sequential Organ Failure Assessment score
severity of disease classification | 28 days
  acute physiology and chronic health evaluation score
critical care need | 28 days
  days on oxygen supply
inflammatory markers | 28 days
  C-Reactive protein
immune profile | 28 days
  C-Reactive protein
fluid status | 28 days
  albumin
oxygen supply | 28 days
  arterial blood gases

CONTACTS AND LOCATIONS:
Overall Officials: Nada H Farrag, Msc, Study Director — NewGiza University (NGU)- School of Pharmacy
Locations (1):
- NewGizaU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No